CLINICAL TRIAL: NCT07127328
Title: Benefits of an Orthodontic Device (Removable Functional Appliance in the Management of Malocclusions/Orofacial Dysfunctions
Brief Title: Benefits of an Orthodontic Device Removable Functional Appliance in the Management of Malocclusions/Orofacial Dysfunctions
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 25Odonto04
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-07

CONDITIONS: Orthodontic Appliances
MeSH Terms: interventions — Orthodontics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Patient with removable funcitonal appliance — Patients who have a malocclusion and/or a dysfunction treated by removable functional appliance
  Other Names: orthodontic treatment

SUMMARY:
The removable functional appliance's goal is to restore functional balance (breathing, swallowing, chewing, etc.) and muscular balance (facial muscles, etc.) in the child. This promotes the establishment of a harmonious and stable occlusion.. The objective of this study is to investigate the benefits of an orthodontic device (removable functional appliance ) in the management of malocclusions/orofacial dysfunctions

ELIGIBILITY:
Inclusion Criteria:

* Patients who had a malocclusion and/or a dysfunction which can be treated by removable functionnal appliance

Exclusion Criteria:

* Patients who don't need a removable functionnal appliance.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who had a malocclusion and/or a dysfunction which can be treated by removable functionnal appliance.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Improvment of malocclusion dysfunctions with removable functional appliances | A follow-up every 6 weeks for 6 months.
  The improvment of malocclusion is evaluated with the observation of photography and videos with cephalometric analyze (Steiner).
Correction of dysfunctions with removable functional appliances | A follow-up every 6 weeks for 6 months.
  The correction is evaluated with the observation of photography and videos with cephalometric analyze (Steiner).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU NICE, Nice, Alpes Maritimes, France